CLINICAL TRIAL: NCT02184780
Title: Impact of Perinatal Anaesthesia and Analgesia on Neurocognitive Outcomes in Early Childhood (PANO Study)
Brief Title: Impact of Perinatal Anaesthesia and Analgesia on Neurocognitive Outcomes in Early Childhood
Acronym: PANO
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: Institute for Human Development and Potential (IHDP), Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: CIRB/2013/644/D
Record Dates: First submitted 2014-07-03; First posted 2014-07-09 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2017-03

CONDITIONS: Anaesthesia; Neurodevelopment
Keywords: Neurodevelopment; General Anaesthesia; Infants; Epidural; Spinal; Anxiety and depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- GUSTO Neurocognitive Cohort: This study involves retrospective analysis of data from an existing cohort of 600 infants who were enrolled in the neurocognitve arm of the GUSTO study (Growing up in Singapore Towards Healthy Outcomes). GUSTO is a prospective observational cohort study done in Singapore, where subjects were followed up from in-utero up to 36 months of age and beyond. The infants have already undergone a rigorous battery of neurocognitive tests at 6, 18, 24 and 36 months of age and their detailed demographic and medical information are available.

SUMMARY:
This study aims to determine the impact of perinatal exposure to anaesthesia and analgesia on neurocognitive outcomes in early childhood by analyzing neurocognitive data already obtained from the local prospective observational cohort study: Growing up in Singapore Towards Healthy Outcomes (GUSTO).

We hypothesize that:

1. Perinatal exposure to anaesthesia and analgesia is associated with poorer neurocognitive outcomes at 6, 18, 24 and 36 months.
2. Maternal anxiety and depression during the antenatal and post-partum period is associated with poorer neurocognitive outcomes at 6, 18 24 and 36 months.

DETAILED DESCRIPTION:
Early exposure to general anesthesia is associated long-term neurocognitive and behavioral abnormalities. However the impact of obstetric and perinatal exposure to anaesthesia and analgesia on long term neurocognitive outcomes in the absence of concurrent events (e.g. fetal hypoxia) is unknown. We aim to determine the impact of perinatal exposure to anaesthesia and analgesia on neurocognitive outcomes in early childhood by analyzing information already obtained from the local prospective observational cohort study: Growing up in Singapore Towards Healthy Outcomes (GUSTO). GUSTO is a large prospective cohort trial currently conducted in Singapore examining maternal and neonatal outcomes including metabolic, psychological and developmental outcomes.

Information on infants' neurocognitive outcomes up to 24 months old are already available and we will correlate these outcomes to

1. The infants' perinatal exposure to anaesthesia and analgesia, as obtained from hospital records, and
2. Maternal anxiety and depression, as observed from analysis of questionnaires already available from GUSTO.

We hypothesize that:

1. Perinatal exposure to anaesthesia and analgesia is associated with poorer neurocognitive outcomes at 6, 18, 24 and 36 months.
2. Maternal anxiety and depression during the antenatal and post-partum period is associated with poorer neurocognitive outcomes at 6, 18 24 and 36 months.

ELIGIBILITY:
Inclusion Criteria:

Infants who are enrolled in the neurocognitve arm of the GUSTO study (Growing up in Singapore Towards Healthy Outcomes).

Exclusion Criteria:

No information available on previous exposure (maternal exposure in utero, perinatal and postnatal exposure) to general anaesthesia, spinal or epidural anaesthesia.

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study involves retrospective analysis of data from an existing cohort of 600 infants who were enrolled in the neurocognitve arm of the GUSTO study (Growing up in Singapore Towards Healthy Outcomes). GUSTO is a prospective observational cohort study done in Singapore, where subjects were followed up from in-utero up to 36 months of age and beyond. The infants have already undergone a rigorous battery of neurocognitive tests at 6, 18, 24 and 36 months of age and their detailed demographic and medical information are available.
Sampling Method: Non-Probability Sample
Enrollment: 468 (Estimated)
Dates: Start 2013-09; Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive score | 24 months of age
  Composite Bayley-III Scores in the following domains tested at 24 months of age (cognitive, language, motor, socio-emotional, general adaptability) These scores are already available from the existing cohort and will be correlated with perinatal exposure to anaesthesia and analgesia and maternal anxiety and depression.

SECONDARY OUTCOMES:
Neurocognitive Score (Deferred Imitation) | 6, 18 and 24 months
  Neurocognitive scores as measured by deferred imitation, a test of memory and attention. These scores are already available from the existing cohort and will be correlated with perinatal exposure to anaesthesia and analgesia and maternal anxiety and depression.

CONTACTS AND LOCATIONS:
Overall Officials: Choon L Bong, MBChB, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore